CLINICAL TRIAL: NCT01073956
Title: Efficacy of Electrotherapy in Subacromial Impingement Syndrome: Randomised Placebo-controlled Clinical Trial
Brief Title: Efficacy of Electrotherapy in Subacromial Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio Espai Salut (Other)
Collaborators: Corporación Fisiogestión S.A. (Unknown); Hospital Clinic of Barcelona (Other); Agència d'Avaluació de Tecnologia i Recerca Mèdiques (Other)
Responsible Party: Conxita Closa Rusinés, Corporación Fisiogestión
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: FES-2009-01
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Subacromial Impingement Syndrome; Shoulder Pain; Physical therapy; Electrotherapy; Ultrasonic therapy; Medium-wave 448 kHz therapy
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Inactive electrotherapy (Placebo Comparator): Inactive electrotherapy is applied to the painful points
  Interventions: Procedure: Inactive electrotherapy
- Ultrasound (Active Comparator): Ultrasound electrotherapy is applied to the painful points
  Interventions: Procedure: Ultrasonic therapy
- Monopolar radiofrequency (Active Comparator): Monopolar radiofrequency electrotherapy is applied to the painful points
  Interventions: Procedure: Medium-wave 448 kHz therapy

INTERVENTIONS:
Procedure: Medium-wave 448 kHz therapy — 0.5 MHz radiofrequency for 10 minutes. At SPS insertion and bicipital groove
  Other Names: Monopolar radiofrequency
  Arms: Monopolar radiofrequency
Procedure: Ultrasonic therapy — Pulsed 1 MHz ultrasound at 2 W/cm2 for 10 minutes. At SPS insertion and bicipital-groove
  Other Names: Ultrasound electrotherapy
  Arms: Ultrasound
Procedure: Inactive electrotherapy — Inactive electrotherapy, inactive head, dosage 0 W/cm2 for 10 minutes. At SPS insertion and bicipital groove.
  Arms: Inactive electrotherapy

SUMMARY:
The purpose of this study is to determine the efficacy of electrotherapy as a coadjuvant in mobility and exercise treatment in the reduction of pain intensity in subacromial impingement syndrome.

DETAILED DESCRIPTION:
Among the different diagnoses covered by the concept of shoulder pain, the most common is subacromial impingement syndrome, which represents 44%-60% of the total.Specific supervised exercises obtain improvements in the range of movement and muscular function by restoring the shoulder's mobility and stability. Physiotherapeutic options include several electrotherapy techniques.

Ultrasound is no more beneficial than exercise alone. Likewise, the results of some more recent studies evaluating the application of ultrasound alone versus placebo, showed that ultrasound alone in physiotherapy treatment of shoulder pain is only effective in patients with calcific tendonitis of the shoulder. All the authors, however, suggest that effectiveness can vary, depending on application conditions, dosage and timing.

The primary objective of the trial is to analyze the efficacy of electrotherapy treatment (monopolar radiofrequency or ultrasound) coadjuvant to mobility and exercise therapy in the reduction of pain intensity in subacromial impingement syndrome.

The secondary objectives of this study are to determine the differences between three intervention groups: monopolar radiofrequency, ultrasound and inactive radiofrequency, in improvement of performance status, quality of life and global impression of improvement.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Shoulder pain secondary to subacromial impingement syndrome
* Pain at rest and/or with free movement and/or with movement against resistance with a score on the visual analogue scale of 3 or higher.
* Documented X-ray (XR), ultrasound (US) and/or magnetic resonance imaging (MRI) evidence of cuff injury involving oedema, tendonitis, fibrosis or torn tendon.
* Potentially available for the next six months.

Exclusion Criteria:

* Documented US and/or MRI evidence of complete tearing of the cuff and clinical inability to lift the arm (drop arm sign)
* Radiological findings of tumour lesions, avascular necrosis, glenoid development defects, acromial bone, severe degenerative signs affecting inter-articular space and fractures
* Limited range of passive movement with capsular pattern
* Recent history of trauma (contusion, falls or sudden jarring)
* Ischaemic cardiopathy in subacute phase
* History of more than five infiltrations and/or shoulder surgery
* History of rehabilitation treatment for the same reason in the last 12 months
* Cognitive deficit, psychiatric alterations or behavioural disorders that might compromise the patient's collaboration
* Unsuitable for electrotherapy: pregnancy, epilepsy, pacemaker, osteosynthesis, undergoing treatment with Sintrom
* Patients in litigation or in the process of making work-related claims
* Failure to understand Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Variation of pain intensity | 12 sessions (1 month)
  Evaluation after 12 sessions of intervention (1 month)

SECONDARY OUTCOMES:
Variation at pain intensity | 18 sessions (1.5 months)
  Evaluation at 1.5 months
Variation at pain intensity | 6 months after intervention
  Follow-up evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Conxita Closa, MD, Principal Investigator — Corporación Fisiogestión S.A.
Locations (2):
- Spain (2):
  - Instituto de Rehabilitación Tres Torres -IR3T, Barcelona, Barcelona
  - Centro de Recuperación Funcional (CRF), Barcelona, Barcelona

REFERENCES:
- [Background] Green S, Buchbinder R, Hetrick S. Physiotherapy interventions for shoulder pain. Cochrane Database Syst Rev. 2003;2003(2):CD004258. doi: 10.1002/14651858.CD004258. PMID 12804509